CLINICAL TRIAL: NCT04325256
Title: Accuracy of Different Scoring Systems for Predicting Successful Induction of Labor: a Cross-sectional Study
Brief Title: Accuracy of Different Scoring Systems for Predicting Successful Induction of Labor
Status: Completed | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Ahmed Mohamed Abbas, Principal investigator, Assiut University
Other Study IDs: IOLSC
Record Dates: First submitted 2020-03-26; First posted 2020-03-27 (Actual); Last update posted 2022-08-25 (Actual); Status verified 2022-08

CONDITIONS: Induction of Labor Affected Fetus / Newborn

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- study group: All pregnant women who will attend the labor unit for induction of labour due to different indications during the study period will be invited to participate in the study.
  Interventions: Procedure: Manipal ultrasound scoring system; Procedure: Levine scoring system

INTERVENTIONS:
Procedure: Manipal ultrasound scoring system — length of the cervix from the internal to external os, presence or absence of funneling and if present width and length of funneling at internal os were measured. Distance between presenting part to external os will be measured and position of the cervix i.e. whether curved or straight will also noted.
Procedure: Levine scoring system — maternal height, parity, body-mass index (BMI) at delivery and the results of modified Bishop's score in calculation of probability of CS

SUMMARY:
Induction of labour (IOL) nowadays is a common procedure in obstetric practice. Presently, IOL is done for 20% of pregnancies for various maternal and fetal indications and nearly 20% of labour inductions end up in caesarean deliveries. The success of IOL mainly depends upon "favourability" of the cervix which is usually assessed by manual examination and Scored as Bishop Score. However, this method is limited by subjectivity and reproducibility and though done in all the patients prior to IOL, several studies have demonstrated poor correlation between Bishop Score and outcome of IOL

ELIGIBILITY:
Inclusion Criteria:

1. Singleton pregnancy.
2. Pregnant ≥ 37 weeks gestation.
3. Fetus with longitudinal lie and vertex presentation.
4. Intact membranes.
5. No vaginal bleeding.

Exclusion Criteria:

1. Patients with previous cesarean delivery.
2. Previous uterine surgery.
3. Antepartum hemorrhage.
4. Cephalopelvic disproportion.
5. Category II or III non-stress test.
6. Malpresentation.
7. Intrauterine fetal death.
8. Fetal growth restriction.
9. Fetuses with major congenital malformations

Sex: Female
Age Groups: Child, Adult, Older Adult
Study Population: pregnant women who will attend the labor unit for induction
Sampling Method: Probability Sample
Enrollment: 400 (Actual)
Dates: Start 2020-12-01 (Actual); Primary Completion 2022-05-31 (Actual); Study Completion 2022-07-15 (Actual)

PRIMARY OUTCOMES:
The rate of successful induction of labor | 24 hours
  an ability to achieve the active phase of labor corresponding to a cervical dilatation of ≥4 cm within 12 h of initiating oxytocin on the first day of induction

CONTACTS AND LOCATIONS:
Locations (1):
- Ahmed Abbas, Assiut, Cairo Governorate, Egypt